CLINICAL TRIAL: NCT04672993
Title: Exploratory Study of a New Urine Collection Device for Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP326
Record Dates: First submitted 2020-09-03; First posted 2020-12-17 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urine Collection Device for Men (Experimental): Test of Urine Collection Device for Men for 7 (+/- 3/0 days).
  Interventions: Device: Urine collection device for men

INTERVENTIONS:
Device: Urine collection device for men — Use of urine collection device for men

SUMMARY:
The aim of the investigation is to evaluate the subjects experience of a new collection device for men.

An open-labelled, single arm study design was chosen for this investigation with a duration of 1 week + up to 3 days extra.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Male
3. Be at least 18 years of age and have full le-gal capacity
4. Suffering from urinary incontinence equiva-lent to using up to 6 pads or 2 diapers per day
5. Have had current incontinence issues for at least 3 months
6. Able to understand patient information and able to change the product himself
7. Up to 6 of the subjects can be users who are using an intermittent catheter due to re-tention, but who are also dribble inconti-nent in-between catheterizations, and hence need a product to handle the inconti-nence.
8. Able to fit the test product.

Exclusion Criteria:

1. If experiencing incontinence less than once per week
2. Bedridden, using wheelchair or using a walking aids regularly

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rasmussen, Principal Investigator
Locations (1):
- Flying Nurses, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no pre-assignment period.
Period: Overall Study
Arm/Group | Urine Collection Device for Men
Started | 20
Completed | 20 (20 participants completed the trial, but data from one participant was lost.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Urine Collection Device for Men
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Found the Product to be Comfortable to Wear
Description: Questionnaire used to measure the frequency of success in support of "comfortable": "How comfortable was the product to wear?". The question was asked at the end of the trial.
Time Frame: One week
Population: ITT (electronic data from one subject was lost)
Measure: Number (95% Confidence Interval); unit: percentages of participants
Arm/Group | Urine Collection Device for Men
Number analyzed (Participants) | 19
percentages of participants | 53 [29 to 76]

ADVERSE EVENTS:
Time Frame: 1 week
Description: Definition of adverse events are from ISO Standard 14155:2021.
  Collection of AEs happened during the 1 week trial and when the subjects terminated their participations by the study nurse and by use of specific forms.
Arm/Group | Urine Collection Device for Men
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urine Collection Device for Men (N=20)
mild skin irritation (Skin and subcutaneous tissue disorders) | 10 (10) — Red and sore skin.
Mild pain (Skin and subcutaneous tissue disorders) | 3 (3) — Pain in the area of the product

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT04672993/Prot_SAP_000.pdf